CLINICAL TRIAL: NCT03807947
Title: Radial Versus Femoral Access for Superselective Embolization of Hepatocellular Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Humanitas Clinical and Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICHRadialTAE
Record Dates: First submitted 2018-12-25; First posted 2019-01-17 (Actual); Last update posted 2019-01-17 (Actual); Status verified 2019-01

CONDITIONS: Hepatocellular Carcinoma; Hepatocellular Carcinoma Non-resectable
Keywords: embolisation, therapeutic; Embolization, Therapeutic; Hepatocellular Carcinoma; HCC; TAE
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radial access (Experimental)
  Interventions: Procedure: Radial TAE - Bland embolization with 40-100 Microparticles
- Transfemoral Access (Active Comparator)
  Interventions: Procedure: Transfemoral TAE - Bland embolization with 40-100 Microparticles

INTERVENTIONS:
Procedure: Radial TAE - Bland embolization with 40-100 Microparticles — TAE - Bland embolization with 40-100 Microparticles performed via left transradial access
  Arms: Radial access
Procedure: Transfemoral TAE - Bland embolization with 40-100 Microparticles — TAE - Bland embolization with 40-100 Microparticles performed via right transfemoral access
  Arms: Transfemoral Access

SUMMARY:
The aim of this prospective, randomized study is to compare TRA vs TFA for superselective embolization of HCC using bland microparticles performed by multiple operators.

In particular, main objectives are to compare:

1. the success rates of TRA and TFA including crossing over events between techniques
2. the inter-operator outcomes in terms of time to complete the vascular access and the vessel catheterization
3. access-related adverse events
4. patient preference and reported discomfort

DETAILED DESCRIPTION:
Hepatic arterial chemoembolization is a safe, proven, and effective technique for the treatment of a number of malignancies, including primary and secondary tumors [1, 2]. This endovascular treatment is performed via femoral artery access in most cases. In the last decades, the transradial approach (TRA) has emerged as a valid alternative to the transfemoral approach (TFA), and it is commonly used in coronary angioplasty as well as stent placement. In particular, shorter monitoring time after the procedure, earlier ambulation, shorter hospital stay and less discomfort associated with potentially reduced bleeding risks make TRA an attractive alternative to TFA.

To date, only one study exists comparing TRA vs TFA in liver embolizations [3]. However, it is non-randomized and reports only the outcomes of one operator performing lobar embolization for multiple liver malignancies.

The aim of this prospective, randomized study is to compare TRA vs TFA for superselective embolization of HCC using bland microparticles performed by multiple operators.

In particular, main objectives are to compare:

1. the success rates of TRA and TFA including crossing over events between techniques
2. the inter-operator outcomes in terms of time to complete the vascular access and the vessel catheterization
3. access-related adverse events
4. patient preference and reported discomfort

ELIGIBILITY:
Inclusion criteria:

* patients affected by HCC with indication to TAE from a multidisciplinary team discussion.

Exclusion criteria

* TAE for other malignancies or bleedings;
* Pregnancy.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2019-01 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Pain and discomfort during and after procedures | 24 hours after intervention
  Questionnaire with four questions with 5 a points scale describing pain and discomfort during and after procedure, where 0 is the minimum and 4 the maximum.

SECONDARY OUTCOMES:
Access-related adverse events | 0-48h after intervention.
  Complication at the site of access like hematoma or pseudoaneurysm

CONTACTS AND LOCATIONS:
Overall Officials: EZIO LANZA, MD, Principal Investigator — Humanitas Research Hospital IRCCS, Rozzano-Milan
Locations (1):
- Humanitas Research Hospital, Rozzano, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Iezzi R, Pompili M, Posa A, Annicchiarico E, Garcovich M, Merlino B, Rodolfino E, Di Noia V, Basso M, Cassano A, Barone C, Gasbarrini A, Manfredi R, Colosimo C. Transradial versus Transfemoral Access for Hepatic Chemoembolization: Intrapatient Prospective Single-Center Study. J Vasc Interv Radiol. 2017 Sep;28(9):1234-1239. doi: 10.1016/j.jvir.2017.06.022. Epub 2017 Jul 27. PMID 28757286